CLINICAL TRIAL: NCT00788515
Title: Comparison of the Safety and Efficacy of Volinanserin and Lormetazepam in the Treatment of Insomnia Characterized by Sleep Maintenance Difficulties. A 4 Week,Randomized, Double-blind, Comparative, Parallel-group Study.
Brief Title: Comparison of Volinanserin and Lormetazepam in the Treatment of Insomnia Characterized by Sleep Maintenance Difficulties
Acronym: REST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision due to absence of demonstration of efficacy of volinanserin in primary insomnia with predominant sleep maintenance problems
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10550; EudraCT: 2008-001492-30
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: insomnia; sleep maintenance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — volinanserin; lormetazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Volinanserin (M100907)
- 2 (Active Comparator)
  Interventions: Drug: Lormetazepam

INTERVENTIONS:
Drug: Volinanserin (M100907) — 2 mg tablets QD
  Arms: 1
Drug: Lormetazepam — 1 mg tablets (overencapsulated) QD
  Arms: 2

SUMMARY:
The primary objective is to compare the potential for next-day residual effects of volinanserin 2 mg/day and lormetazepam 1 mg/day by measuring the sleepiness in the morning using the patient's sleep questionnaire during 4 weeks of treatment in patients with chronic primary insomnia and sleep maintenance difficulties.

Secondary objectives are to compare the clinical safety of both products, including the potential for rebound insomnia and withdrawal symptoms after treatment discontinuation, to compare the efficacy of both products on subjective sleep parameters and to compare the effects of both products on patient's daytime functioning.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients with Primary Insomnia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria

Exclusion Criteria:

* Based on patient's information, the patient has spent less than 6.5 hours or more than 9.0 hours, in bed, each night, over the preceding two weeks
* Based on patient's information, the patient complains of less than one hour of wakefulness after sleep onset for at least 3 nights per week over the preceding month
* Disturbances of sleep maintenance parameters based on the patient's sleep questionnaire during the run-in period differing from pre-defined criteria.
* Pregnant or breastfeeding women and women of childbearing potential without effective contraceptive method of birth control
* Night shift workers and individuals who nap 3 or more times per week
* Consumption of xanthine-containing beverages (i.e., tea, coffee or cola) that comprises more than 5 cups or glasses per day

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Sleepiness in the morning measured on a visual analog scale of the patient's sleep questionnaire | 4 weeks

SECONDARY OUTCOMES:
Other measure of next-day residual effects (ability to concentrate of the patient's sleep questionnaire) | 4 weeks
Rebound effect measured by pr-WASO and pr-SOL on patient's sleep questionnaire during the run-out period | 4 weeks
Subjective sleep parameters | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden